CLINICAL TRIAL: NCT06374108
Title: Effects of Supervised Progressive Resistance Training on Central Nervous System Functioning (Corticospinal Excitability) and Walking Capacity in Persons With Multiple Sclerosis
Brief Title: Resistance Training and Corticospinal Excitability in Multiple Sclerosis
Acronym: NEXIMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Neuro_Exercise
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose resistance training (Active Comparator): 10 weeks intervention with 2.5 weekly supervised resistance training sessions (2 or 3 sessions/week for high dose resistance training; 25 sessions in total).
  Interventions: Behavioral: Progressive resistance training
- Low dose resistance training (Active Comparator): 10 weeks intervention with 1 weekly supervised resistance training session (low dose resistance training; 10 sessions in total).
  Interventions: Behavioral: Progressive resistance training
- Waitlist control. (No Intervention): The waitlist control group will initially be instructed to maintain their normal daily activity during the 10 week intervention period. Hereafter, they will be offered a 10 week high dose resistance training intervention that combines supervised and home based exercise sessions .

INTERVENTIONS:
Behavioral: Progressive resistance training — The RT exercise regime will focus on lower extremity exercises (60-90% of 1 repetition maximum) as well as incorporating functional exercises.
  Arms: High dose resistance training; Low dose resistance training

SUMMARY:
The goal of the present study is to investigate effects of progressive resistance training on central nervous system functioning (corticospinal excitability (CSE)) and walking capacity in persons with multiple sclerosis (pwMS). A total of 54 pwMS will be enrolled and randomized into 1 of 3 groups: high dose resistant training (RT), low dose RT, and waitlist control.

DETAILED DESCRIPTION:
Neurodegeneration is a hallmark of multiple sclerosis (MS), affecting both structure and function of the central nervous system (CNS). Neurodegeneration is the main driver of disability progression in MS, evidenced by studies showing deleterious structural and functional CNS changes, ultimately reducing quality of life. Consequently, the interaction between the nervous system and muscular system undergoes deleterious changes causing reduced neuromuscular function (i.e., ability to develop muscle strength and power) and physical function.

The functional CNS changes have been evidenced by using the non invasive brain stimulation technique Transcranial Magnetic Stimulation, showing decreased corticospinal excitability alongside increased central motor conduction time. Moreover, functional peripheral nervous system (PNS) changes have been evidenced by nerve conduction methods, revealing decreased amplitude of compound muscle action potential and increased latency of nerve signaling. In an ongoing exploratory study (unpublished), the investigators have observed that functional CNS and PNS outcomes deteriorate with disability progression from healthy to mildly to moderately disabled people with MS (PwMS).

Exercise is beneficial from both an individual and a societal perspective, and has proven to be both safe and without any noticeable side effects in PwMS. Resistance training (RT) appears particularly effective in improving neuromuscular function (mainly muscle strength) and physical function (especially walking capacity). Whilst RT and other exercise modalities may elicit positive effects on CNS structure in PwMS, it seems to require a long-term (≥ 6 months) exposure. In contrast, CNS (and potentially PNS) function may adapt much more rapidly, despite a scarcity of studies (and with heterogeneous findings) involving PwMS. Interestingly, an exploratory exercise study (non-controlled, low sample size, 10 weeks treadmill walking intervention) assessed corticospinal excitability in PwMS, and observed substantial improvements after the intervention. Apart from this study, a major knowledge gap exists in terms of elucidating the potential beneficial effects of exercise (RT in particular) on CNS (and PNS) function. Based on evidence from healthy young individuals, substantial improvements in corticospinal excitability have been shown following 2-12 weeks of RT, supporting that RT-induced improvements in corticospinal excitability can also be seen in PwMS. Lastly, as existing exercise guidelines for PwMS fails to refer to evidence on dose-response to exercise, and a recent systematic review on exercise studies found no dose-response studies in PwMS (n=202), this aspect is also of great clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* MS diagnosis according to the McDonald diagnostic criteria
* Shows impairments in walking capacity
* Ability to self transport to test and exercise

Exclusion Criteria:

* Pregnancy
* Neurological or other comorbidities that affects the nervous system
* Relapse within the past 2 months
* Pacemaker or metallic implants
* Hypertension (medically unregulated)
* Participation in structured RT over the past 3 months (≥ 2 sessions/week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
MEP/Mmax ratio | Change from Baseline to 10 weeks
  Cortical excitability measured as amplitude percentage ratio between MEP (resting) and Mmax (Cmap of TA). Unit (intended): %

SECONDARY OUTCOMES:
Muscle strength | Change from Baseline to 10 weeks
  Maximal voluntary contraction (MVC) is the maximal force-generating capacity (plantar flexion and dorsal flexion). Unit (intended): N
Voluntary activation I | Change from Baseline to 10 weeks
  Assessed by Interpolated Twitch Technique (ITT) (dorsal flexion). Unit (intended): %
Voluntary activation II | Change from Baseline to 10 weeks
  EMG amplitude during MVC (plantar flexion and dorsal flexion). Unit (intended): μV
Force Steadiness | Change from Baseline to 10 weeks
  A quantitative measure of the ability to control muscle tonus (dorsal flexion). Unit (intended): root-mean-square (RMS) error (Coefficient of Variation (CV))
Rate of Force Developement | Change from Baseline to 10 weeks
  This is defined as the speed at which the contractile elements of the muscle can develop force (plantar flexion and dorsal flexion). Unit (intended): N/s
Ultrasound | Change from Baseline to 10 weeks
  Measure of muscle thickness of the tibialis anterior. Unit (intended): mm
Resting Motor Threshold (rMT) | Change from Baseline to 10 weeks
  The intensity necessary to produce a motor-evoked potential (MEP) that exceeds a defined peak-to-peak amplitude (50 μV) 50% of the time in a finite number of trials. Unit (intended): % Maximum stimulator output (MSO)
Active Motor Threshold (aMT) | Change from Baseline to 10 weeks
  The intensity necessary to produce a motor-evoked potential (MEP) that exceeds a defined peak-to-peak amplitude (50 μV) 50% of the time in a finite number of trials during voluntary activation (20% of MVC). Unit (intended): % Maximum stimulator output (MSO)
MEP latency (resting) | Change from Baseline to 10 weeks
  The transmission time from stimulating the cortex to the start of the evoked potential in the EMG of the target muscle. Unit (intended): ms
MEP latency (active) | Change from Baseline to 10 weeks
  The transmission time from stimulating the cortex to the start of the evoked potential in the EMG of the target muscle. Unit (intended): ms
MEP amplitude (resting) | Change from Baseline to 10 weeks
  Peak-to-peak of averaged MEP (20 stimulations of 120% rMT). Unit (intended): mV
MEP amplitude (active) | Change from Baseline to 10 weeks
  Peak-to-peak of averaged MEP (20 stimulations of 120% rMT). Unit (intended): mV
Short-interval intracortical Inhibition (SICI) | Change from Baseline to 10 weeks
  SICI measures cortical inhibition and is a TMS protocol in which two stimuli are delivered with an interstimulus interval (ISI) of 2.5 ms. Unit (intended): the relative amplitude difference of motor evoked potentials (MEPs) (%).
Intracortical facilitation (ICF) | Change from Baseline to 10 weeks
  ICF measures cortical facilitation and is a TMS protocol in which two stimuli are delivered with an interstimulus interval (ISI) of 10 ms. Unit (intended): the relative amplitude reduction of motor evoked potentials (MEPs) (%).
Cortical Silent Period (CSP) | Change from Baseline to 10 weeks
  The temporary interruption of electromyographic signal from a muscle following a motor-evoked potential (MEP) triggered by transcranial magnetic stimulation (TMS). Unit (intended): ms
Central Motor Conduction Time (CMCT) | Change from Baseline to 10 weeks
  The time it takes for the fastest action potentials to travel from the site of cortical stimulation to the spinal motoneuron. It is calculated by subtracting the peripheral motor conduction time (PMCT) from the MEP latency or by the F-wave method. Unit (intended): ms
EEG-EMG coherence (0-1) | Change from Baseline to 10 weeks
  Synchronization between brain activity (EEG) and muscle activity (EMG) over a specific frequency range. Unit (intended): ranging from 0 to 1, where 0 is no coherence and 1 is perfect coherence.
Timed 25 feet walk test (T25FWT) | Change from Baseline to 10 weeks
  Objective test that measures walking speed. Unit (intended): seconds.
6-minute walk test (6MWT) | Change from Baseline to 10 weeks
  Objective test that measures walking endurance. Unit (intended): meters.
Six spot step test (SSST) | Change from Baseline to 10 weeks
  Objective test that measures walking coordination and balance. Unit (intended): seconds.
5 sit-to-stand (5STS) | Change from Baseline to 10 weeks
  Objective test that measures functional lower limb muscle strength and power. Unit (intended): seconds.
9-step stair ascend (9SSA) | Change from Baseline to 10 weeks
  Objective test that measures functional lower limb muscle strength and power. Unit (intended): seconds.
Patient determined disease steps (PDDS) | Change from Baseline to 10 weeks
  A patient-reported measure of disability. Unit (intended): score (0-8; 0 is normal).
Multiple Sclerosis Walking Scale (MSWS) | Change from Baseline to 10 weeks
  Questionnaire that measures quality of life. Unit (intended): score (0-100; 0 is better).
Modified fatigue impact scale (MFIS) | Change from Baseline to 10 weeks
  Questionnaire that measures the impact fatigue has on daily life. Unit (intended): score (0-84; 0 is better)
MS impact scale (MSIS) | Change from Baseline to 10 weeks
  Questionnaire that measures the impact MS has on daily life. Unit (intended): score (29-145; 29 is better)
Falls-efficacy scale - international (FES-1) | Change from Baseline to 10 weeks
  Questionnaire that measures concerns about falling. Unit (intended): score (16-64; 16 is better)
The Physical Activity Enjoyment Scale (PACES) | Change from Baseline to 10 weeks
  Questionnaire that measures enjoyment for physical activity. Unit (intended): score (8-56; Higher score reflect greater level of enjoyment)
Brief pain inventory (BPI) | Change from Baseline to 10 weeks
  Questionnaire that measures pain severity and pain interference. Unit (intended): No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
Baecke physical activity | Change from Baseline to 10 weeks
  Questionnaire (patient-reported outcome) assessing patient-reported participation in physical activities. Unit (intended): Score range is continuous (0-xx). Higher is better.
Accelerometry | Change from Baseline to 10 weeks
  Method used to measures and analyze movement and acceleration in three dimensions of a person (physical activity). Unit (intended): g (m/s^2)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Public Health, Aarhus, Central Jutland
  - Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Copenhagen N